CLINICAL TRIAL: NCT04781036
Title: The Study of Foot-skin Microbiome and Metabolomics of Thai Naval Cadets With Pitted Keratolysis
Brief Title: Foot-skin Microbiome and Metabolomics of Pitted Keratolysis
Acronym: Foot-skin M&M
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Charussri Leeyaphan, Associate Professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PK microbiome and metabolomic
Record Dates: First submitted 2021-02-25; First posted 2021-03-04 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Microbial Disease; Metabolomics
Keywords: Pitted keratolysis; Microbiome; Metabolomics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Normal feet (No Intervention): * Swab their feet to analyze foot microbiome via 16s DNA sequencing
  * Collect their socks to analyze metabolomics via gas chromatography
- Foot odor without pitted keratolysis (Experimental): * Swab their feet to analyze foot microbiome via 16s DNA sequencing
  * Collect their socks to analyze metabolomics via gas chromatography
  * Apply 4% chlorhexidine for 2 weeks
  * Re-evaluate their feet at time of treatment finish and 1 months after treatment finish. The forementioned methods (swab and collect their socks) will be applied on their feet again.
  * The microbiome and metabolomics will be analyzed to evaluate the difference of microbe and substances after treatment.
  Interventions: Drug: 4%Chlorhexidine
- Foot odor with pitted keratolysis (Experimental): * Swab their feet to analyze foot microbiome via 16s DNA sequencing
  * Collect their socks to analyze metabolomics via gas chromatography
  * Apply 4% chlorhexidine for 2 weeks
  * Re-evaluate their feet at time of treatment finish and 1 months after treatment finish. The forementioned methods (swab and collect their socks) will be applied on their feet again.
  * The microbiome and metabolomics will be analyzed to evaluate the difference of microbe and substances after treatment.
  Interventions: Drug: 4%Chlorhexidine

INTERVENTIONS:
Drug: 4%Chlorhexidine — 4%Chlorhexidine was given to participants with foot odor for 2 weeks
  Arms: Foot odor with pitted keratolysis; Foot odor without pitted keratolysis

SUMMARY:
This study aimed to investigate the skin microbiome and metabolomics of patients with pitted keratolysis.

DETAILED DESCRIPTION:
Pitted keratolysis is a skin infectious disease which can cause an unpleasant smell that can affect self-confidence and interpersonal relationships. The research problem was initiated through a community outreach program organized by the Department of Dermatology Siriraj Hospital, Thailand. From many years of experiences, our dermatologist teams observed that pitted keratolysis was a common disease among naval cadets who wore enclosed footwear for long hours, and it was more prevalent after a boot camp that spanned over months. This disease is chronic with no efficient standard treatment and limited information on the pathogenesis of the disease. Therefore, we propose to conduct a study on the pathogenesis of pitted keratolysis and malodorous feet through a longitudinal study of foot-skin microbiome and associated volatile metabolomic profiles of foot odor. With the unique population, with similar age range, daily activities, and diet, this study will allow to focus on the association of changes in microbiome in relation to pathogenesis of pitted keratolysis and malodorous feet, with fewer cofounding factors.

The skin microbiome is a group of various microorganisms, such as bacteria, fungi, and viruses, residing on skin. Human skin microbiome can differ with respect to age, ethnicity, diet, climate and environment. Recently, there have been numerous studies highlighting the association of microbes with pathogenesis of various skin diseases, such as atopic dermatitis, acne vulgaris, and psoriasis (references?). In this project, we hypothesize that the alteration of skin microbiome as well as changes in metabolite profiles can be associated with the mechanism of the disease. The skin microbiome data generated in this study will be analyzed for microbial profiles using the QIIME2, a next-generation microbiome bioinformatics platform, and a graphic software package, "Statistical Analysis of Taxonomic and Functional Profiles" (STAMP). In parallel, we will apply a high throughput gas chromatography mass-spectrometry-based metabolomics to detect volatile metabolites present in foot odor in association with the observed foot-skin microbiome. This metabolite information will not only provide an additional aspect of pathogenesis of the disease but also might offer a new standard indicator of foot odor that can be further used in clinical practice. Finally, skin microbiome and metabolomic data will be analyzed using various methods of correlation analysis as well as integrative analysis to gain deeper understanding of the disease mechanism at the molecular levels.

The outcomes of this project will provide insights into the pathogenesis of pitted keratolysis. The scientific knowledge gained from the study will be translated into a more effective treatment of the disease. The human microbiome of healthy population and the disease-specific microbiome data will lay the groundwork to develop a human microbiome database for Thai people. Additionally, the success of the project will allow the development of advanced instrumental methodology and an integrative analysis approach to analyze multi -omics data, which will be great assets in advancing multidisciplinary research.

ELIGIBILITY:
Inclusion Criteria:

* Naval rating cadets at Chumpol Naval Rating School, Thailand who volunteer to participate in this study. Informed consent will be obtained from all participants.
* Age ≥ 18 years.
* No underlying disease.
* Normal BMI (18.5-22.9 kg/m2).
* No previous history of pitted keratolysis.
* No previous history of dermatophytosis complex.
* Refrain from washing their feet for 12 hours prior to sampling.

Exclusion Criteria:

* Volunteers who have taken medication or topical antibiotics for pitted keratolysis within 2 weeks before the enrollment.
* Volunteers who have taken oral antibiotics within 2 weeks before enrollment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Amount of skin microbiome | 2 months
  Foot-skin microbial profiles of healthy Thai people and patients with pitted keratolysis
Composition of microbiota at skin | 2 months
  Foot-skin microbial profiles of healthy Thai people and patients with pitted keratolysis

SECONDARY OUTCOMES:
Amount of metabolite in foot odor | 2 months
  Metabolite profiling of foot odor

CONTACTS AND LOCATIONS:
Overall Officials: Sumanas Bunyaratavej, MD, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Department of Dermatology Siriraj Hospital, Bangkoknoi, Bangkok
  - Department of Dermatology Siriraj Hospital, Bangkok

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Grice EA, Segre JA. The skin microbiome. Nat Rev Microbiol. 2011 Apr;9(4):244-53. doi: 10.1038/nrmicro2537. PMID 21407241
- [Background] Musthaq S, Mazuy A, Jakus J. The microbiome in dermatology. Clin Dermatol. 2018 May-Jun;36(3):390-398. doi: 10.1016/j.clindermatol.2018.03.012. Epub 2018 Mar 10. PMID 29908581
- [Background] Perez Perez GI, Gao Z, Jourdain R, Ramirez J, Gany F, Clavaud C, Demaude J, Breton L, Blaser MJ. Body Site Is a More Determinant Factor than Human Population Diversity in the Healthy Skin Microbiome. PLoS One. 2016 Apr 18;11(4):e0151990. doi: 10.1371/journal.pone.0151990. eCollection 2016. PMID 27088867
- [Background] Sander MA, Sander MS, Isaac-Renton JL, Croxen MA. The Cutaneous Microbiome: Implications for Dermatology Practice. J Cutan Med Surg. 2019 Jul/Aug;23(4):436-441. doi: 10.1177/1203475419839939. Epub 2019 Apr 2. PMID 30938174
- [Background] Yu Y, Dunaway S, Champer J, Kim J, Alikhan A. Changing our microbiome: probiotics in dermatology. Br J Dermatol. 2020 Jan;182(1):39-46. doi: 10.1111/bjd.18088. Epub 2019 Jul 28. PMID 31049923
- [Background] Szabo K, Erdei L, Bolla BS, Tax G, Biro T, Kemeny L. Factors shaping the composition of the cutaneous microbiota. Br J Dermatol. 2017 Feb;176(2):344-351. doi: 10.1111/bjd.14967. Epub 2017 Jan 23. PMID 27518483
- [Background] Schoch JJ, Monir RL, Satcher KG, Harris J, Triplett E, Neu J. The infantile cutaneous microbiome: A review. Pediatr Dermatol. 2019 Sep;36(5):574-580. doi: 10.1111/pde.13870. Epub 2019 Jul 23. PMID 31332846
- [Background] Iebba V, Totino V, Gagliardi A, Santangelo F, Cacciotti F, Trancassini M, Mancini C, Cicerone C, Corazziari E, Pantanella F, Schippa S. Eubiosis and dysbiosis: the two sides of the microbiota. New Microbiol. 2016 Jan;39(1):1-12. PMID 26922981
- [Background] Thomas CL, Fernandez-Penas P. The microbiome and atopic eczema: More than skin deep. Australas J Dermatol. 2017 Feb;58(1):18-24. doi: 10.1111/ajd.12435. Epub 2016 Jan 28. PMID 26821151
- [Background] Holmes E, Wilson ID, Nicholson JK. Metabolic phenotyping in health and disease. Cell. 2008 Sep 5;134(5):714-7. doi: 10.1016/j.cell.2008.08.026. PMID 18775301
- [Background] Patti GJ, Yanes O, Siuzdak G. Innovation: Metabolomics: the apogee of the omics trilogy. Nat Rev Mol Cell Biol. 2012 Mar 22;13(4):263-9. doi: 10.1038/nrm3314. PMID 22436749
- [Background] Melnik BC. Linking diet to acne metabolomics, inflammation, and comedogenesis: an update. Clin Cosmet Investig Dermatol. 2015 Jul 15;8:371-88. doi: 10.2147/CCID.S69135. eCollection 2015. PMID 26203267
- [Background] Nordstrom KM, McGinley KJ, Cappiello L, Zechman JM, Leyden JJ. Pitted keratolysis. The role of Micrococcus sedentarius. Arch Dermatol. 1987 Oct;123(10):1320-5. doi: 10.1001/archderm.123.10.1320. PMID 3310909
- [Background] Singh G, Naik CL. Pitted keratolysis. Indian J Dermatol Venereol Leprol. 2005 May-Jun;71(3):213-5. doi: 10.4103/0378-6323.16250. No abstract available. PMID 16394424
- [Background] Bolyen E, Rideout JR, Dillon MR, Bokulich NA, Abnet CC, Al-Ghalith GA, Alexander H, Alm EJ, Arumugam M, Asnicar F, Bai Y, Bisanz JE, Bittinger K, Brejnrod A, Brislawn CJ, Brown CT, Callahan BJ, Caraballo-Rodriguez AM, Chase J, Cope EK, Da Silva R, Diener C, Dorrestein PC, Douglas GM, Durall DM, Duvallet C, Edwardson CF, Ernst M, Estaki M, Fouquier J, Gauglitz JM, Gibbons SM, Gibson DL, Gonzalez A, Gorlick K, Guo J, Hillmann B, Holmes S, Holste H, Huttenhower C, Huttley GA, Janssen S, Jarmusch AK, Jiang L, Kaehler BD, Kang KB, Keefe CR, Keim P, Kelley ST, Knights D, Koester I, Kosciolek T, Kreps J, Langille MGI, Lee J, Ley R, Liu YX, Loftfield E, Lozupone C, Maher M, Marotz C, Martin BD, McDonald D, McIver LJ, Melnik AV, Metcalf JL, Morgan SC, Morton JT, Naimey AT, Navas-Molina JA, Nothias LF, Orchanian SB, Pearson T, Peoples SL, Petras D, Preuss ML, Pruesse E, Rasmussen LB, Rivers A, Robeson MS 2nd, Rosenthal P, Segata N, Shaffer M, Shiffer A, Sinha R, Song SJ, Spear JR, Swafford AD, Thompson LR, Torres PJ, Trinh P, Tripathi A, Turnbaugh PJ, Ul-Hasan S, van der Hooft JJJ, Vargas F, Vazquez-Baeza Y, Vogtmann E, von Hippel M, Walters W, Wan Y, Wang M, Warren J, Weber KC, Williamson CHD, Willis AD, Xu ZZ, Zaneveld JR, Zhang Y, Zhu Q, Knight R, Caporaso JG. Author Correction: Reproducible, interactive, scalable and extensible microbiome data science using QIIME 2. Nat Biotechnol. 2019 Sep;37(9):1091. doi: 10.1038/s41587-019-0252-6. PMID 31399723
- [Result] Li M, Budding AE, van der Lugt-Degen M, Du-Thumm L, Vandeven M, Fan A. The influence of age, gender and race/ethnicity on the composition of the human axillary microbiome. Int J Cosmet Sci. 2019 Aug;41(4):371-377. doi: 10.1111/ics.12549. PMID 31190339
- [Result] Zhu T, Liu X, Kong FQ, Duan YY, Yee AL, Kim M, Galzote C, Gilbert JA, Quan ZX. Age and Mothers: Potent Influences of Children's Skin Microbiota. J Invest Dermatol. 2019 Dec;139(12):2497-2505.e6. doi: 10.1016/j.jid.2019.05.018. Epub 2019 Aug 13. PMID 31420081
- [Result] Shami A, Al-Mijalli S, Pongchaikul P, Al-Barrag A, AbduRahim S. The prevalence of the culturable human skin aerobic bacteria in Riyadh, Saudi Arabia. BMC Microbiol. 2019 Aug 16;19(1):189. doi: 10.1186/s12866-019-1569-5. PMID 31419942
- [Result] Blaser MJ, Dominguez-Bello MG, Contreras M, Magris M, Hidalgo G, Estrada I, Gao Z, Clemente JC, Costello EK, Knight R. Distinct cutaneous bacterial assemblages in a sampling of South American Amerindians and US residents. ISME J. 2013 Jan;7(1):85-95. doi: 10.1038/ismej.2012.81. Epub 2012 Aug 16. PMID 22895161
- [Result] Kong HH, Oh J, Deming C, Conlan S, Grice EA, Beatson MA, Nomicos E, Polley EC, Komarow HD; NISC Comparative Sequence Program; Murray PR, Turner ML, Segre JA. Temporal shifts in the skin microbiome associated with disease flares and treatment in children with atopic dermatitis. Genome Res. 2012 May;22(5):850-9. doi: 10.1101/gr.131029.111. Epub 2012 Feb 6. PMID 22310478
- [Result] Tsilochristou O, du Toit G, Sayre PH, Roberts G, Lawson K, Sever ML, Bahnson HT, Radulovic S, Basting M, Plaut M, Lack G; Immune Tolerance Network Learning Early About Peanut Allergy Study Team. Association of Staphylococcus aureus colonization with food allergy occurs independently of eczema severity. J Allergy Clin Immunol. 2019 Aug;144(2):494-503. doi: 10.1016/j.jaci.2019.04.025. Epub 2019 May 31. PMID 31160034
- [Result] Zheng Y, Wang Q, Ma L, Chen Y, Gao Y, Zhang G, Cui S, Liang H, He C, Song L. Alterations in the skin microbiome are associated with disease severity and treatment in the perioral zone of the skin of infants with atopic dermatitis. Eur J Clin Microbiol Infect Dis. 2019 Sep;38(9):1677-1685. doi: 10.1007/s10096-019-03598-9. Epub 2019 May 31. PMID 31152265
- [Result] Quan C, Chen XY, Li X, Xue F, Chen LH, Liu N, Wang B, Wang LQ, Wang XP, Yang H, Zheng J. Psoriatic lesions are characterized by higher bacterial load and imbalance between Cutibacterium and Corynebacterium. J Am Acad Dermatol. 2020 Apr;82(4):955-961. doi: 10.1016/j.jaad.2019.06.024. Epub 2019 Jun 19. PMID 31228520
- [Result] Dutkiewicz EP, Hsieh KT, Wang YS, Chiu HY, Urban PL. Hydrogel Micropatch and Mass Spectrometry-Assisted Screening for Psoriasis-Related Skin Metabolites. Clin Chem. 2016 Aug;62(8):1120-8. doi: 10.1373/clinchem.2016.256396. Epub 2016 Jun 20. PMID 27324733
- [Result] Sitter B, Johnsson MK, Halgunset J, Bathen TF. Metabolic changes in psoriatic skin under topical corticosteroid treatment. BMC Dermatol. 2013 Aug 14;13:8. doi: 10.1186/1471-5945-13-8. PMID 23945194
- [Result] Yan D, Afifi L, Jeon C, Trivedi M, Chang HW, Lee K, Liao W. The metabolomics of psoriatic disease. Psoriasis (Auckl). 2017;7:1-15. doi: 10.2147/PTT.S118348. Epub 2017 Jan 31. PMID 28824870
- [Result] Longshaw CM, Wright JD, Farrell AM, Holland KT. Kytococcus sedentarius, the organism associated with pitted keratolysis, produces two keratin-degrading enzymes. J Appl Microbiol. 2002;93(5):810-6. doi: 10.1046/j.1365-2672.2002.01742.x. PMID 12392527
- [Result] Woodgyer AJ, Baxter M, Rush-Munro FM, Brown J, Kaplan W. Isolation of Dermatophilus congolensis from two New Zealand cases of pitted keratolysis. Australas J Dermatol. 1985 Apr;26(1):29-35. doi: 10.1111/j.1440-0960.1985.tb01811.x. No abstract available. PMID 4062746
- [Result] Svejgaard E, Christophersen J, Jelsdorf HM. Tinea pedis and erythrasma in Danish recruits. Clinical signs, prevalence, incidence, and correlation to atopy. J Am Acad Dermatol. 1986 Jun;14(6):993-9. doi: 10.1016/s0190-9622(86)70122-9. PMID 3722494
- [Result] Bunyaratavej S, Leeyaphan C, Chanyachailert P, Pattanaprichakul P, Ongsri P, Kulthanan K. Clinical manifestations, risk factors and quality of life in patients with pitted keratolysis: a cross-sectional study in cadets. Br J Dermatol. 2018 Nov;179(5):1220-1221. doi: 10.1111/bjd.16923. Epub 2018 Sep 14. No abstract available. PMID 29951993
- [Result] Kaptanoglu AF, Yuksel O, Ozyurt S. Plantar pitted keratolysis: a study from non-risk groups. Dermatol Reports. 2012 Feb 7;4(1):e4. doi: 10.4081/dr.2012.e4. eCollection 2012 Jan 2. PMID 25386314
- [Result] Makhecha M, Dass S, Singh T, Gandhi R, Yadav T, Rathod D. Pitted keratolysis - a study of various clinical manifestations. Int J Dermatol. 2017 Nov;56(11):1154-1160. doi: 10.1111/ijd.13744. Epub 2017 Sep 18. PMID 28924971
- [Result] Takama H, Tamada Y, Yano K, Nitta Y, Ikeya T. Pitted keratolysis: clinical manifestations in 53 cases. Br J Dermatol. 1997 Aug;137(2):282-5. doi: 10.1046/j.1365-2133.1997.18211899.x. PMID 9292083
- [Result] Leeyaphan C, Bunyaratavej S, Taychakhoonavudh S, Kulthanachairojana N, Pattanaprichakul P, Chanyachailert P, Ongsri P, Arunkajohnsak S, Limphoka P, Kulthanan K. Cost-effectiveness analysis and safety of erythromycin 4% gel and 4% chlorhexidine scrub for pitted keratolysis treatment. J Dermatolog Treat. 2019 Sep;30(6):627-629. doi: 10.1080/09546634.2018.1543846. Epub 2018 Dec 11. PMID 30415588
- [Result] Leung MH, Wilkins D, Lee PK. Insights into the pan-microbiome: skin microbial communities of Chinese individuals differ from other racial groups. Sci Rep. 2015 Jul 16;5:11845. doi: 10.1038/srep11845. PMID 26177982